CLINICAL TRIAL: NCT02399514
Title: Verbesserung Der Schlafqualität Durch RePneu® Coils Zur Behandlung Des Fortgeschrittenen Lungenemphysems
Brief Title: Improvement of Sleep Quality by RePneu® Coils in Advanced Pulmonary Emphysema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Principal Investigator, Karl Josef Franke, Senior Physician, Helios Klinik Ambrock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JF001 sleep
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: COPD; Emphysema
Keywords: Sleep; emphysema; coils; lung volume reduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RePneum coils (Other): Patients who needed lung volume reduction with RePneum coils
  Interventions: Other: Polysomnographic diagnostic

INTERVENTIONS:
Other: Polysomnographic diagnostic — Polysomnographic diagnostic performed one prior to Coil Treatment, one six months after and one twelve month after Coil Treatment
  Other Names: PSG

SUMMARY:
Improvement of sleep quality in emphysema patients is desirable. Yet, there are no data of patients treated with RePneu coils. This monocenter prospective study investigates the effect on sleep quality of RePneu coils for reduction of dynamic hyperinflation in advanced disease stages of pulmonary emphysema.

Patient's sleep will be studied in three Polysomnography measurement nights, one prior to Coil Treatment, one six months after, and one twelve month after.

Primary objective is to investigate differences in sleep quality 6 and 12 months after Coil Treatment.

Further endpoints are changes in daily activity and sleep (actigraphy), 6MWT, lung function parameters, and questionnaires (SGRQ, mMRC dyspnoe scale).

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* RePneu Coil treatment according to clinical criteria

Exclusion Criteria:

* Pregnancy or nursing period
* Participation in another clinical trial within the last 4 weeks
* Incapable of giving consent
* Known OSA (AHI>10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency, measured in baseline and 6 and 12 month after coil treatment. | 3 times in one year
  Sleep Efficiency is evaluated by the ratio of WASO (Time "wake after sleep onset") to Sleep Period Time (SPT).

SECONDARY OUTCOMES:
Quality of life Questionnaire | 3 times in one year
  The St. George Respiratory Questionnaire (SGRQ) is designed to capture the health related quality of life.

OTHER OUTCOMES:
Activity: Physical activity measured by an actimeter over 7 days, before and 6 month after the coil treatment. The device is able to capture activity levels, sleep and wake times . | 1 week in baseline and 6 month after coil treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Josef Franke, MD, Principal Investigator — Helios Klinik Ambrock
Locations (1):
- Helios Klinik Ambrock, Hagen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Franke KJ, Domanski U, Schroder M, Nilius G. Effects of endobronchial coils for endoscopic lung volume reduction on sleep in COPD patients with advanced pulmonary emphysema. Sleep Breath. 2021 Jun;25(2):727-735. doi: 10.1007/s11325-020-02176-0. Epub 2020 Aug 26. PMID 32845475